CLINICAL TRIAL: NCT01142388
Title: Randomized Phase II Study of Paclitaxel With or Without the Anti-IGF-IR mAb Cixutumumab (IMC-A12) as Second Line Treatment for Patients With Metastatic Esophageal or GE Junction Cancer
Brief Title: Paclitaxel With or Without Cixutumumab as Second-Line Therapy in Treating Patients With Metastatic Esophageal Cancer or Gastroesophageal Junction Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02045; NCI-2011-02045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E2208; CDR0000674327; E2208 (Other: ECOG-ACRIN Cancer Research Group); E2208 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Esophageal Adenocarcinoma; Metastatic Esophageal Squamous Cell Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Recurrent Esophageal Adenocarcinoma; Recurrent Esophageal Carcinoma; Recurrent Esophageal Squamous Cell Carcinoma; Recurrent Gastroesophageal Junction Adenocarcinoma; Stage IV Esophageal Cancer AJCC v7
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — cixutumumab; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study
- Arm II (cixutumumab, paclitaxel) (Experimental): Patients receive cixutumumab IV over 1 hour on days 1 and 15, and paclitaxel as in Arm I.
  Interventions: Biological: Cixutumumab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC A12; IMC-A12; IMCA12
  Arms: Arm II (cixutumumab, paclitaxel)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial studies how well paclitaxel with or without cixutumumab works in treating patients with esophageal cancer or gastroesophageal junction cancer that has spread to other places in the body (metastatic). Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cixutumumab may kill cancer cells by blocking the action of a protein needed for cancer cell growth. Giving paclitaxel with or without cixutumumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival of paclitaxel plus cixutumumab (IMC-A12) versus paclitaxel alone as second-line therapy in patients with metastatic esophagus or gastroesophageal (GE) junction cancer.

SECONDARY OBJECTIVES:

I. To evaluate the overall survival of paclitaxel plus cixutumumab (IMC-A12) versus paclitaxel alone in this patient population.

II. To evaluate the response rate of paclitaxel plus cixutumumab (IMC-A12) versus paclitaxel alone in this patient population.

III. To evaluate the toxicity of cixutumumab (IMC-A12) plus paclitaxel versus paclitaxel alone in this patient population.

IV. Exploratory analyses will assess potentially relevant cixutumumab (IMC-A12) pharmacodynamic biomarkers obtained from serum samples, including but not limited to, insulin-like growth factor (IGF)-I, IGF-II, insulin-like growth factor binding protein (IGFBP)-2, and IGFBP-3.

OUTLINE: Patients are equally randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 1 hour at a dose of 80 mg/m^2 on days 1, 8, and 15 of every 28 day cycle.

ARM II: Patients receive cixutumumab IV over 1 hour at a dose of 10 mg/kg on days 1 and 15 of every 28 day cycle and paclitaxel as in Arm I.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy >= 12 weeks
* Women must not be pregnant or breast-feeding due to potential harm to fetus from cixutumumab (IMC-A12) and paclitaxel; all females of childbearing potential must have a blood test or urine study within 48 hours prior to registration to rule out pregnancy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method or birth control; abstinence) for the duration of study therapy and for 3 months after the last dose of cixutumumab (IMC-A12); should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have measurable disease
* Patients must have metastatic disease of the esophagus or gastroesophageal junction

  * Histologic, cytologic or radiologic documentation of metastatic squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction; radiologic, endoscopic, histologic or cytologic evidence of locally recurrent or locally residual (post-resection) disease is also permitted
  * For the purposes of this study, undifferentiated adenocarcinomas and adenosquamous tumors will be considered as adenocarcinomas; in addition, tumors involving the gastroesophageal junction will be defined by the Siewert classification
* Patients with gastroesophageal junction tumors who are eligible:

  * Adenocarcinoma of the esophageal junction (AEG) Type I: adenocarcinoma of the distal esophagus which usually arises from an area with specialized intestinal metaplasia of the esophagus, i.e., Barrett's esophagus, and may infiltrate the esophagogastric junction from above
  * AEG Type II: true carcinoma of the cardia arising from the cardiac epithelium or short segments with intestinal metaplasia at the esophagogastric junction
* Patients with gastroesophageal junction tumors who are NOT eligible:

  * AEG Type III: subcardial gastric carcinoma which infiltrates the esophagogastric junction and distal esophagus from below
* Patients must have received and progressed on one and only one line of prior systemic therapy for esophagus or esophagogastric cancer; this could have included one regimen for metastatic disease, or one regimen with radiotherapy for initially locally advanced disease; prior radiation therapy is permitted

  * If patients progress or recur within 6 months of neoadjuvant/adjuvant therapy, this will be considered one line of therapy; for patients progressing or recurring more than 6 months after neoadjuvant/adjuvant therapy, they will need to receive one line of therapy for recurrent disease to be eligible
  * If patients receive one regimen in which a chemotherapy agent is dropped for toxicity without progression, this treatment will be considered one line of therapy; however, substitution or addition of a new agent will be considered a second line of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Leukocytes > 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine transaminase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional ULN
* Creatinine =< 1.5 X institutional ULN or creatinine clearance >= 60 mL/min/1.73m^2 for patients with creatinine levels above institutional normal
* Patients must have fasting serum glucose =< 160 mg/dL (8.8 mmol/L) or =< ULN, and hemoglobin A1C =< 7% (0.07 International System of Units [SI units]) within 14 days of registration; if baseline nonfasting glucose =< 160 mg/dL (8.8 mmol/L), fasting glucose measurement is not required
* Registration no fewer than 28 days from last chemotherapy
* A "currently active" second malignancy other than non-melanoma skin cancers are not to be registered; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse

Exclusion Criteria:

* Patients have received prior taxane or anti-insulin growth factor receptor (IGFR) therapy
* Patients must not have any of the following conditions:

  * Poorly controlled diabetes mellitus; patients with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range (fasting glucose =< 160 mg/dL [8.8 mmol/L] or below the ULN and hemoglobin A1C =< 7% [0.07 SI units]) and that they are on a stable dietary or therapeutic regimen for this condition
  * Recent major surgery, hormonal therapy (other than replacement) or chemotherapy, within 4 weeks prior to entering the study or those who have not recovered from adverse events
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to cixutumumab (IMC-A12)
  * Psychiatric illness that would prevent the patient from giving informed consent
* Medical conditions such as active/uncontrolled infection (including HIV) or cardiac disease that would make this protocol unreasonably hazardous for the patient in the opinion of the treating physician; cardiac disease may include uncontrolled high blood pressure, unstable angina, or serious uncontrolled cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-09-21 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Cohen, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (233):
- United States (233):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Trinity Medical Center, Moline, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Stockton S, Catalano P, Cohen SJ, Burtness BA, Mitchell EP, Dotan E, Lubner SJ, Kumar P, Mulcahy MF, Fisher GA, Crandall TL, Benson A. Paclitaxel With or Without Cixutumumab as Second-Line Treatment of Metastatic Esophageal or Gastroesophageal Junction Cancer: A Randomized Phase II ECOG-ACRIN Trial. Oncologist. 2023 Sep 7;28(9):827-e822. doi: 10.1093/oncolo/oyad096. PMID 37104870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on September 21, 2010 and closed to accrual on October 15, 2012 with total accrual of 94 patients from 27 ECOG-ACRIN affiliated institutions.
Groups:
- Arm I (Paclitaxel): Patients receive paclitaxel IV over 1 hour at a dose of 80 mg/m^2 on days 1, 8, and 15 of every 28 day cycle.
  paclitaxel: Given IV
- Arm II (Cixutumumab, Paclitaxel): Patients receive cixutumumab IV over 1 hour at a dose of 10 mg/kg on days 1 and 15 of every 28 day cycle, and paclitaxel as in Arm I.
  cixutumumab: Given IV, administered prior to chemotherapy, doses were based on actual body weight
  paclitaxel: Given IV
Period: Overall Study
Arm/Group | Arm I (Paclitaxel) | Arm II (Cixutumumab, Paclitaxel)
Started | 47 | 47
Eligible | 43 | 44
Treated | 40 | 44
Completed | 0 (Treatment continued until disease progression or intolerable toxicity.) | 0
Not Completed | 47 | 47
Not completed — Lack of Efficacy | 21 | 31
Not completed — Adverse Event | 9 | 5
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Alternative therapy | 1 | 0
Not completed — Other complications | 0 | 2
Not completed — Other | 1 | 1
Not completed — Never started therapy | 7 | 3

BASELINE CHARACTERISTICS:
Population: Per protocol, the primary population for all efficacy endpoints is all eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel) | Arm II (Cixutumumab, Paclitaxel) | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Median (Full Range); unit: years] | 63 [40 to 89] | 62 [40 to 82] | 62 [40 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 35 | 33 | 68
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from randomization to progression or death without evidence of progression. For cases without documentation of progression, follow-up was censored at the date of last disease assessment without progression, unless death occurred within a short period of time (4 months) following the date last known progression-free, in which case the death was counted as an event, or in the case of death within 4 months of randomization in the absence of disease evaluation before that time. PFS was estimated using the Kaplan-Meier method, with 90% confidence intervals calculated using Greenwood's formula, and compared by the log rank test.
Time Frame: assessed every 3 months for 2 years after registration
Population: Eligible patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel) | Arm II (Cixutumumab, Paclitaxel)
Number analyzed (Participants) | 43 | 44
months | 2.6 [1.8 to 4.1] | 2.3 [2.0 to 3.6]
Statistical Analysis 1: Comparison: Arm I (Paclitaxel) vs Arm II (Cixutumumab, Paclitaxel); Test type: Superiority or Other; p = 0.85, Log Rank; one-sided stratified log rank test, stratifying on: 1) gastroesophageal junction vs. esophagus, 2) squamous cell carcinoma vs. adenocarcinoma

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization until death (event), or censored at last date known alive. OS was estimated using the Kaplan-Meier method, with 90% confidence intervals calculated using Greenwood's formula, and compared by the log rank test.
Time Frame: assessed every 3 months for 2 years after registration
Population: Eligible patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel) | Arm II (Cixutumumab, Paclitaxel)
Number analyzed (Participants) | 43 | 44
months | 6.5 [4.6 to 9.5] | 6.4 [4.9 to 8.0]
Statistical Analysis 1: Comparison: Arm I (Paclitaxel) vs Arm II (Cixutumumab, Paclitaxel); Test type: Superiority or Other; p = 0.50, Log Rank; one-sided stratified log rank test, stratifying on 1) gastroesophageal junction vs. esophagus, 2) squamous cell carcinoma vs. adenocarcinoma

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as number of patients with complete response (CR) or partial response (PR) divided by all eligible patients. Responses are evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level. PR is defined as disappearance of target lesions or at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: assessed every 8 weeks while on treatment and every 3 months after treatment for 2 years
Population: Eligible patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Paclitaxel) | Arm II (Cixutumumab, Paclitaxel)
Number analyzed (Participants) | 43 | 44
percentage of participants | 12 [5 to 23] | 14 [6 to 25]

ADVERSE EVENTS:
Time Frame: Assessed at the end of each cycle (1 cycle=28 days) while on treatment and for 30 days after the end of treatment
Description: Late adverse events (defined as any adverse events that occur prior to diagnosis of progression/relapse and has not been previously reported) are collected via the long-term follow up form at each required follow-up visits.
Arm/Group | Arm I (Paclitaxel) | Arm II (Cixutumumab, Paclitaxel)
Serious Adverse Events (participants affected / at risk) | 21/40 | 23/44
Other Adverse Events (participants affected / at risk) | 39/40 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel) (N=40) | Arm II (Cixutumumab, Paclitaxel) (N=44)
Anemia (Blood and lymphatic system disorders) | 4 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 1
Infusion related reaction (General disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Sepsis (Infections and infestations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 8 | 8
Neutrophil count decreased (Investigations) | 3 | 8
Platelet count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel) (N=40) | Arm II (Cixutumumab, Paclitaxel) (N=44)
Anemia (Blood and lymphatic system disorders) | 29 | 29
Edema limbs (General disorders) | 4 | 1
Fatigue (General disorders) | 27 | 27
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 8 | 10
Mucositis oral (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 8 | 14
Vomiting (Gastrointestinal disorders) | 6 | 9
Alanine aminotransferase increased (Investigations) | 5 | 4
Alkaline phosphatase increased (Investigations) | 5 | 10
Aspartate aminotransferase increased (Investigations) | 5 | 8
Creatinine increased (Investigations) | 0 | 4
Lymphocyte count decreased (Investigations) | 17 | 15
Neutrophil count decreased (Investigations) | 10 | 14
Platelet count decreased (Investigations) | 6 | 10
Weight loss (Investigations) | 8 | 8
White blood cell decreased (Investigations) | 13 | 18
Anorexia (Metabolism and nutrition disorders) | 7 | 12
Glucose intolerance (Metabolism and nutrition disorders) | 3 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 6
Hyponatremia (Metabolism and nutrition disorders) | 3 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 2 | 5
Dysgeusia (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 1 | 4
Paresthesia (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 16
Flashing lights (Eye disorders) | 0 | 7
Floaters (Eye disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less